CLINICAL TRIAL: NCT06536478
Title: The Effect of Exercise Intervention on Posture, Trunk Flexibility and Spine Function in Patients With Parkinson's Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 202307076RIND
Record Dates: First submitted 2024-07-29; First posted 2024-08-05 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2023-09

CONDITIONS: Parkinson Disease
Keywords: Parkinson Disease; exercise; posture
MeSH Terms: conditions — Parkinson Disease; Motor Activity | interventions — Exercise; Educational Status

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- exercise (Experimental): Exercise group will perform 50 minutes of exercise twice a week, including stretching, core exercises, gross motor movements and balance exercises for 5 weeks
  Interventions: Other: exercise
- education (Other): The patient will be given a one-time exercise education session and a 50-minute video that included stretching, core exercises, gross motor movements and balance exercises that could be practiced at home.
  Interventions: Other: education

INTERVENTIONS:
Other: exercise — 50 minutes of exercise twice a week, including stretching, core exercises, gross motor movements and balance exercises for 5 weeks
  Arms: exercise
Other: education — The patient will be given a one-time exercise education session and a 50-minute video that included stretching, core exercises, gross motor movements and balance exercises that could be practiced at home.
  Arms: education

SUMMARY:
The primary goal of this clinical trail is to compare the effect of a five-week specific motor interventions on the postural alignment, trunk range of motion and spine function in patients with Parkinson's disease. The secondary goal is to investigate the effect of specific motor interventions on pain, balance, gait, and quality of life.

Participants will:

be randomly allocated to a control group or an exercise group and will perform 50 minutes of exercise twice a week, including stretching, core exercises, gross motor movements and balance exercises for 5 weeks. Each group will be assessed for posture, trunk range of motion, spine function, pain, balance, gait, and quality of life before and after the intervention.

DETAILED DESCRIPTION:
Participants will be randomly allocated to a control group or an exercise group and will perform 50 minutes of exercise twice a week, including stretching, core exercises, gross motor movements and balance exercises for 5 weeks. Each group will be assessed for posture, trunk range of motion, spine function, pain, balance, gait and quality of life before and after the intervention.

Posture evaluation was performed by measuring the angles of Flexion and Side-bending, by placing marks on the Spinal process of 7th cervical spine and the Spinal process of 5th lumbar spine, and by taking images of the Sagittal plane and Frontal plane. A digital flat-panel camera was used to take images in the sagittal plane and the coronal plane, and the angle between the line connecting the seventh cervical process of the spine and the fifth lumbar process of the lumbar spine and the vertical line was measured on the images; the angle in the coronal plane was defined as the anterior tilt angle, and that in the coronal plane was defined as the lateral bending angle.

Trunk flexion range of motion is measured using a goniometer and a tape measure in the following manner: Trunk flexion range of motion is measured with the trunk flexed anteriorly: the starting position of the case is standing in an upright position, and the tape measure is fixed to the seventh cervical vertebrae and the first vertebrae on the spinous processes, then the case is asked to relax the trunk forward to the end of the flexion without anteriorly tilting the pelvis. The difference between the tape measure in forward bending and upright position was taken as the value of trunk anterior tilt mobility. Trunk extension range of motion: The starting position of the case was standing in an upright position, and a tape measure was fixed on the spinous processes of the seventh cervical vertebrae and the first vertebrae of the recommended vertebrae. After the case was asked to relax the trunk with both hands and bend the trunk back to the bottom without tilting the pelvis posteriorly, and the difference between the posterior bending and the tape measure in the upright position was used as a value of the trunk extension range of motion. Trunk side-bending range of motion: The starting position of the case was standing upright, the center of the joint goniometer was aligned with the spinal process of the first segment of the recommended vertebrae of the case, one side of the goniometer was perpendicular to the floor, and the other side was aligned with the seventh segment of the cervical vertebrae of the case, the case was asked to make a left/right side-bending motion, and the angle between the left/right side-bending and the upright position was subtracted as the value of trunk side-bending range of motion. The angle between the left/right lateral bend and the upright position was subtracted to obtain the value of trunk lateral bending activity. Trunk rotation range of motion: With the case in a seated but not reclined position, the center of the joint goniometer was aligned with the center of the case's head, with one side of the goniometer parallel to the line of the iliac crest of the pelvis, and the other side parallel to the line of the shoulder crests on both sides. One side of the goniometer was parallel to the line of the iliac crest of the pelvis and the other side was parallel to the line of the shoulder crests on both sides of the body. The case was asked to perform a left/right rotation, and the angle between the left/right rotation and the seated position was subtracted to obtain a value for the degree of torso rotation.

Spinal function is assessed by evaluating the functional activities related to the spine, including Functional axial rotation and Supine to and from standing. The Functional Axial Rotation Test is performed by asking the patient to use a Cervical Range of Motion (CROM) device in a sitting position to measure the angle of rotation of the case when viewed from the left/right side. The lying to standing test is performed by asking the patient to use a Cervical Range of Motion (CROM) device to measure the angle of rotation of the case when viewed from the right/left side. The Lying to Standing Test measures the time taken by the case to move from standing to lying and lying to standing.

Pain was assessed using the Visual Analogue Scale , VAS, which asks the patient about the degree of low back pain.

The Shortened Version of the Balance Evaluation Systems Tests (Mini-BEST) is used to evaluate balance in cases of balance impairment (e.g., Parkinson's disease, brain injury, vestibular disorders, stroke, or multiple sclerosis). The assessment consists of four sub-balance systems with 14 items each scored 0, 1, or 2 depending on performance, ranging from 0 to 28, with higher scores indicating better balance. The four sub-balance systems included in the test are Anticipatory postural adjustments, Reactive postural control, Sensory orientation and Dynamic gait.

Walking speed was assessed using the 10 m walk test, which involves walking a distance of 14 meters at a comfortable speed and recording the time taken from the second to the twelfth meter in order to calculate the walking speed of the case, with the use of a walking aid if necessary.

The gait assessment will record the parameters of walking and assess them using the Tinetti Mobility Test (TMT). The TMT is used to assess the gait performance of elderly people, people with Parkinson's disease, brain injury, stroke or multiple sclerosis. The assessment is performed by asking the patient to walk a distance of 25 feet in a straight line at a comfortable speed. The administrator can either directly observe or video-record the gait of the patient, or use a walking aid if necessary. The assessment includes the observation of hesitancy to start walking, height of the raised foot, gait length, gait symmetry, continuity of stride, walking path, trunk stability, and width of stride, with a score of 0, 1, or 2 for each item. Each item was scored as 0, 1 or 2, ranging from 0 to 12, with higher scores indicating a more problem-free gait.

Quality of life is assessed using the short version of the Parkinson's Disease Questionnaire (PDQ-8). The PDQ8 is a self-completion questionnaire with eight questions covering eight domains, including activities of daily living, exercise, cognition, social support, communication, emotional well-being, shame, and feelings of physical discomfort, with the lower the score, the better the quality of life and health.

ELIGIBILITY:
Inclusion Criteria:

* Hoehn-Yahr classification 2 to 3
* Regular compliance with medication program
* Stable medical condition and vital signs, conscious
* Be able to follow instructions.

Exclusion Criteria:

* Cognitive impairment or dementia who are unable to cooperate with therapy or functional assessment
* Patients with musculoskeletal injuries or surgeries that have resulted in limited mobility
* Patients with physician-diagnosed cardiorespiratory disorders with activity limitations
* Patients with acute neurological disorders.

Ages: 30 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 40 (Estimated)
Dates: Start 2023-09-28 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
postural alignment of frontal and sagittal plance | before and immediately after the intervention
  The angles of Flexion and Side-bending of the trunk in degrees
range of motion of trunk flexion and side-bending | before and immediately after the intervention
  The range of motion of trunk flexion and side-bending will be evaluated in degrees
Supine to and from sitting | before and immediately after the intervention
  The time of supine to and from sitting is measured in seconds

SECONDARY OUTCOMES:
Visual Analogue Scale of low back pain | before and immediately after the intervention
  It is a scale from 0 to 10. The higher score means the patient has more severe pain.
The Shortened Version of the Balance Evaluation Systems Tests (Mini-BEST) | before and immediately after the intervention
  It is a scale from 0 to 28. The higher score means the patient has no impairment in their balance.
10 meter gait speed | before and immediately after the intervention
  the speed of gait is measured in meters per second
Tinetti Mobility Test (TMT) | before and immediately after the intervention
  It is a scale from 0 to 12. The higher score means the patient has a better gait pattern.
the short version of the Parkinson's Disease Questionnaire (PDQ-8) | before and immediately after the intervention
  quality of life will be measured by the PDQ-8. It is a scale from 0-32. The higher scale means the patient has worse quality of life.
Falls Efficacy Scale International (FES-I) | before and immediately after the intervention
  It is a scale from 16 to 64. The higher score means the patient is more afraid of falling down.

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital Hsinchu Branch, Hsinchu, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Barone P, Santangelo G, Amboni M, Pellecchia MT, Vitale C. Pisa syndrome in Parkinson's disease and parkinsonism: clinical features, pathophysiology, and treatment. Lancet Neurol. 2016 Sep;15(10):1063-74. doi: 10.1016/S1474-4422(16)30173-9. Epub 2016 Aug 8. PMID 27571158
- [Result] Norkin, C.C. and D.J. White, Measurement of Joint Motion: A Guide to Goniometry. 5th ed. 2017: F.A.Davis.
- [Result] Vaugoyeau M, Viallet F, Aurenty R, Assaiante C, Mesure S, Massion J. Axial rotation in Parkinson's disease. J Neurol Neurosurg Psychiatry. 2006 Jul;77(7):815-21. doi: 10.1136/jnnp.2004.050666. Epub 2006 Mar 30. PMID 16574736
- [Result] Schenkman M, Cutson TM, Kuchibhatla M, Chandler J, Pieper CF, Ray L, Laub KC. Exercise to improve spinal flexibility and function for people with Parkinson's disease: a randomized, controlled trial. J Am Geriatr Soc. 1998 Oct;46(10):1207-16. doi: 10.1111/j.1532-5415.1998.tb04535.x. PMID 9777901
- [Result] Delgado DA, Lambert BS, Boutris N, McCulloch PC, Robbins AB, Moreno MR, Harris JD. Validation of Digital Visual Analog Scale Pain Scoring With a Traditional Paper-based Visual Analog Scale in Adults. J Am Acad Orthop Surg Glob Res Rev. 2018 Mar 23;2(3):e088. doi: 10.5435/JAAOSGlobal-D-17-00088. eCollection 2018 Mar. PMID 30211382
- [Result] Duncan RP, Leddy AL, Cavanaugh JT, Dibble LE, Ellis TD, Ford MP, Foreman KB, Earhart GM. Comparative utility of the BESTest, mini-BESTest, and brief-BESTest for predicting falls in individuals with Parkinson disease: a cohort study. Phys Ther. 2013 Apr;93(4):542-50. doi: 10.2522/ptj.20120302. Epub 2012 Nov 21. PMID 23174567
- [Result] Lindholm B, Nilsson MH, Hansson O, Hagell P. The clinical significance of 10-m walk test standardizations in Parkinson's disease. J Neurol. 2018 Aug;265(8):1829-1835. doi: 10.1007/s00415-018-8921-9. Epub 2018 Jun 6. PMID 29876762
- [Result] Kegelmeyer DA, Kloos AD, Thomas KM, Kostyk SK. Reliability and validity of the Tinetti Mobility Test for individuals with Parkinson disease. Phys Ther. 2007 Oct;87(10):1369-78. doi: 10.2522/ptj.20070007. Epub 2007 Aug 7. PMID 17684089
- [Result] Peto V, Jenkinson C, Fitzpatrick R. PDQ-39: a review of the development, validation and application of a Parkinson's disease quality of life questionnaire and its associated measures. J Neurol. 1998 May;245 Suppl 1:S10-4. doi: 10.1007/pl00007730. PMID 9617716